CLINICAL TRIAL: NCT01295008
Title: Androgenetic Alopecia in Fabry Disease
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 010-308
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Male pattern baldness; Alopecia; GLA gene mutation; Alpha-galactosidase A
MeSH Terms: conditions — Fabry Disease; Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with the classic form
- Fabry disease and healthy controls

SUMMARY:
The purpose of this study is to assess whether patients with the classic form of Fabry disease have significantly less androgenic alopecia (male pattern baldness).

DETAILED DESCRIPTION:
Objectives: To test the hypothesis that adult males with classic form of Fabry disease have a significantly lower incidence of androgenic alopecia than matched controls.

Study Population: 120 patients aged 20-64 with Fabry disease that have GLA mutations or alpha-galactosidase A activity associated with no residual enzyme activity and non-Fabry male controls of the same age range and the same number of non-Fabry controls.

Design: This is a cross-sectional study comparing the prevalence of androgenic alopecia in two groups of subjects.

Outcome Measures: The levels of the outcome will be no androgenic alopecia and frontal only androgenetic alopecia opposed to vertex only and frontal and vertex androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with Fabry disease age 20-64 years old.
* Healthy male controls age 20-64 years old
* GLA gene mutations associated with the classic form of Fabry disease or having alpha-galactosidase A activity that is essentially zero
* Patients who freely agree to participate in this study and understand the nature, risks and benefits of this study and give their written informed consent.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Selected from specialy clinic
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2010-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
No and frontal only androgenetic alopecia | 1 Year
  No and frontal only androgenetic alopecia opposed to vertex only and frontal and vertex androgenetic alopecia.

SECONDARY OUTCOMES:
Vertex only and frontal and vertex androgenetic alopecia. | 1 Year
  No and frontal only androgenetic alopecia opposed to vertex only and frontal and vertex androgenetic alopecia.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Schiffmann, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States